CLINICAL TRIAL: NCT01138098
Title: Antibody Persistence and Immune Memory Against the Hepatitis B Antigen in 11-12 Year Old Children, Previously Vaccinated With DTPa-HBV-IPV/Hib Vaccine in Study 217744/031
Brief Title: Evaluation of Antibody Persistence and Immune Memory Against the Hepatitis B Antigen in Previously Vaccinated Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113954
Record Dates: First submitted 2010-05-27; First posted 2010-06-07 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis B
Keywords: Persistence; challenge dose; Engerix-B; immune response
MeSH Terms: conditions — Hepatitis B

ARMS (2):
- Infanrix-hexa/Engerix-B Group (Experimental): Subjects aged 11-12 year old received 3 doses of Infanrix-hexa vaccine in the primary study (217744/031 (NCT01457495)) and a challenge dose of Engerix-B vaccine in this study. Engerix-B was administered as a single dose intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Engerix™-B
- Infanrix-IPV+Hib/Engerix-B Group (Active Comparator): Subjects aged 11-12 year old received 3 doses of Infanrix-IPV+Hib and Engerix-B vaccines in the primary study (217744/031 (NCT01457495)) and a challenge dose of Engerix-B vaccine in this study. Engerix-B was administered as a single dose intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: Engerix™-B — Intramuscular, single dose

SUMMARY:
This study will evaluate the persistence of immunity to hepatitis B 10 to 11 years after vaccination with Infanrix hexa™ or Engerix™-B and also the ability to mount an immune response to the challenge dose of Engerix™-B.

DETAILED DESCRIPTION:
Subjects who participated in the primary study 217744/031 (NCT01457495) will be invited at the age of 11-12 years to participate in this follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/Legally acceptable representative) can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 11-12 years at the time of study entry (from and including the 11th birthday until and excluding the 13th birthday).
* Written informed consent obtained from the parent or Legally Acceptable Representative of the subject.
* Study procedures will be explained to subjects and depending on their understanding, optional informed assent will be sought at the discretion of the investigator.
* Written informed assent obtained from the subject in addition to the informed consent signed by the parent(s)/ Legally Acceptable Representative (s).
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who have received all three doses of Infanrix hexa or Engerix-B in the primary study 217744/031 (NCT01457495).
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Child in care.
* Use of any investigational or non-registered product drug or vaccine) other than the study vaccine within 30 days preceding the challenge dose of HBV vaccine, or planned use during the study period.
* Receipt of hepatitis B (containing) vaccine after vaccination in the primary study 217744/031 (NCT01457495).
* History of hepatitis B disease.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 30 days after the HBV vaccine challenge dose.
* Administration of immunoglobulins and/or any blood products within the three months preceding the challenge dose of HBV vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the challenge dose of HBV vaccine.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Known hypersensitivity to any component of the HBV vaccine or evidence of hypersensitivity after previous immunisation with a vaccine containing the hepatitis B component.
* Acute disease and/or fever at the time of enrolment.
* Fever is defined as temperature ≥ 37.5°C (99.5°F) on oral, axillary or tympanic setting
* Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2010-06-07; Primary Completion 2010-11-26 (Actual); Study Completion 2010-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Slovakia (11):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Dubnica nad Váhom
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nová Dubnica
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Púchov
  - GSK Investigational Site, Rožňava
  - GSK Investigational Site, Trebišov
  - GSK Investigational Site, Zlaté Moravce

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Avdicova M, Crasta PD, Hardt K, Kovac M. Lasting immune memory against hepatitis B following challenge 10-11 years after primary vaccination with either three doses of hexavalent DTPa-HBV-IPV/Hib or monovalent hepatitis B vaccine at 3, 5 and 11-12 months of age. Vaccine. 2015 May 28;33(23):2727-33. doi: 10.1016/j.vaccine.2014.06.070. Epub 2014 Jun 22. PMID 24962750
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Infanrix-hexa/Engerix-B Group: Subjects aged 11-12 year old received 3 doses of Infanrix-hexa vaccine in the primary study (NCT01457495) and a challenge dose of Engerix-B vaccine in this study. Engerix-B was administered as a single dose intramuscularly into the deltoid region of the non-dominant arm.
- Infanrix-IPV+Hib/Engerix-B Group: Subjects aged 11-12 year old received 3 doses of Infanrix-IPV+Hib and Engerix-B vaccines in the primary study (NCT01457495) and a challenge dose of Engerix-B vaccine in this study. Engerix-B was administered as a single dose intramuscularly into the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Started | 95 | 90
Completed | 95 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group | Total
Number analyzed (Participants) | 95 | 90 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.3 (0.46) | 11.3 (0.47) | 11.3 (0.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 80
  Male | 50 | 55 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-hepatitis B (Anti-HBs) Antibody Concentration Equal to or Above (≥) 100 Milli-International Units Per Milliliter (mIU/mL)
Description: A decrease in the specificity of the anti-HB enzyme-linked immunosorbent assay (ELISA) had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: One month after a challenge dose of Engerix-B vaccine
Population: The According-To-Protocol (ATP) cohort for analysis of immunogenicity included all evaluable subjects (i.e. those meeting eligibility criteria, complied with the procedures, with no elimination criteria) who had received a challenge dose Engerix-B vaccine and for whom immunogenicity data were available at the post-Engerix-B challenge time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 94 | 89
Participants | 88 | 84

2. Secondary Outcome: Number of Subjects With an Anamnestic Response to a Challenge Dose
Description: The anamnestic response was defined as: at least (≥) a 4-fold rise in post-challenge dose anti-HBs antibody concentrations in subjects seropositive at the pre-challenge dose time point. - Post-challenge dose anti-HBs antibody concentrations ≥ 10 mIU/mL in seronegative subjects at the pre-challenge dose time point. A seropositive/seronegative subject is a subject with anti-HBs antibody concentration ≥/lower than (<) 6.2 mIU/mL. A decrease in the specificity of the anti-HB ELISA had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis and the initial 3.3 mIU/mL seropositivity cut-off was revised into the new 6.2 mIU/mL cut-off.
Time Frame: Before and one month after a challenge dose of Engerix-B vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 94 | 89
Participants | 91 | 86

3. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentration ≥ 6.2 mIU/mL
Description: A seropositive subject was defined as a subject with anti-HBs antibody concentration ≥ the 6.2 mIU/mLcut-off. A decrease in the specificity of the anti-HB ELISA had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis and the initial 3.3 mIU/mL seropositivity cut-off was revised into the new 6.2 mIU/mL cut-off.
Time Frame: Before and one month after a challenge dose of Engerix-B vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 89
Participants
  ≥ 6.2 mIU/mL [pre-challenge dose] | 53 | 57
  ≥ 6.2 mIU/mL [post-challenge dose]: number analyzed (Participants) | 94 | 89
  ≥ 6.2 mIU/mL [post-challenge dose] | 92 | 88

4. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentration ≥ 10 mIU/mL
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentration ≥ 10 mIU/mL. A decrease in the specificity of the anti-HB enzyme-linked immunosorbent assay (ELISA) had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: Before and one month after a challenge dose of Engerix-B vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 89
Participants
  ≥ 10 mIU/mL [pre-challenge dose] | 46 | 52
  ≥ 10 mIU/mL [post-challenge dose]: number analyzed (Participants) | 94 | 89
  ≥ 10 mIU/mL [post-challenge dose] | 91 | 88

5. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentration ≥ 100 mIU/mL
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentration ≥ 10 mIU/mL. A decrease in the specificity of the anti-HB ELISA had been observed in some studies for low levels of antibody (10-100 mIU/mL). All the available blood samples initially tested with ELISA were re-tested using the Chemi Luminescence Immuno Assay (CLIA) approved by the US Food and Drug Administration (FDA). The table shows updated results following partial or complete retesting/reanalysis.
Time Frame: Before the challenge dose of Engerix-B vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 89
Participants | 14 | 17

6. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling.
Time Frame: During the 4-day (Days 0-3) follow-up period after a challenge dose of Engerix-B vaccine
Population: The Total Vaccinated cohort included all subjects who received the challenge dose of Engerix-B vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 90
Participants
  Pain | 30 | 24
  Redness | 25 | 22
  Swelling | 15 | 8

7. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, gastrointestinal, headache and temperature (Temperature is defined as axillary temparature equal to or above 37.5 degrees Celsius (°C)).
Time Frame: During the 4-day (Days 0-3) follow-up period after a challenge dose of Engerix-B vaccine
Population: The Total Vaccinated cohort included all subjects who received the challenge dose of Engerix-B vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 90
Participants
  Fatigue | 23 | 22
  Gastrointestinal | 9 | 9
  Headache | 19 | 14
  Temperature ≥ 37.5°C | 1 | 3

8. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Days 0-30) follow-up period after a challenge dose of Engerix-B vaccine
Population: The Total Vaccinated cohort included all subjects who received the challenge dose of Engerix-B vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 90
Participants | 5 | 7

9. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: After the challenge dose of Engerix-B vaccine up to the study end
Population: The Total Vaccinated cohort included all subjects who received the challenge dose of Engerix-B vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
Number analyzed (Participants) | 95 | 90
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: During the 4-day (Days 0-3) follow-up period after the challenge dose of Engerix-B vaccine. SAEs: after the challenge dose of Engerix-B vaccine up to the study end
Arm/Group | Infanrix-hexa/Engerix-B Group | Infanrix-IPV+Hib/Engerix-B Group
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/90
Serious Adverse Events (participants affected / at risk) | 1/95 | 0/90
Other Adverse Events (participants affected / at risk) | 48/95 | 43/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-hexa/Engerix-B Group (N=95) | Infanrix-IPV+Hib/Engerix-B Group (N=90)
Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-hexa/Engerix-B Group (N=95) | Infanrix-IPV+Hib/Engerix-B Group (N=90)
Pain (General disorders) | 30 | 24
Redness (General disorders) | 25 | 22
Swelling (General disorders) | 15 | 8
Fatigue (General disorders) | 23 | 22
Gastrointestinal (General disorders) | 9 | 9
Headache (General disorders) | 19 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.